CLINICAL TRIAL: NCT05568758
Title: Effects of Combining Thoracic Lymphatic Pump Technique and Exercises on Patients With Chronic Mechanical Low Back Pain
Brief Title: Thoracic Lymphatic Pump Technique Exercises Chronic Mechanical Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Basma Hesham Hasaneen EL-Fayoumi, physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Thorac lymph exercises back
Record Dates: First submitted 2022-10-01; First posted 2022-10-06 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Low Back Pain, Mechanical
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic lymphatic pump technique (Experimental): The subject lies in the supine position; the therapist stands at the patient's head, facing the subject. The therapist then, places the thenar eminence of each hand to the pectoral region inferior to the clavicle and the other fingers are spread around the thoracic cage and angled toward the body's side to create a consistent, compressive force across the thoracic cage. The subject is then asked to breathe in deeply and breathe out. While breathing out, rhythmic oscillatory compression in the posterior and caudal direction is applied to the chest wall. By the end of the expiratory phase, the compressive force is maintained, and the subject is asked to take another deep breath. In this way, the subject encountered some resistance equivalent to the chest-wall movement during inspiration. The maneuver is repeated for five respiratory cycles, after that the therapist slowly reduces the compressive force and withdraws his hands.
  Interventions: Other: Thoracic lymphatic pump technique; Other: Exercises (stretching and strenghtening )
- exercises (Experimental): Stretching exercises (hamstring stretch-lower back stretch) Strenghening exercises(abdominal curl up-supine bridging-trunk extension)
  Interventions: Other: Exercises (stretching and strenghtening )

INTERVENTIONS:
Other: Thoracic lymphatic pump technique — The subject lies in the supine position; the therapist stands at the patient's head, facing the subject. The therapist then, places the thenar eminence of each hand to the pectoral region inferior to the clavicle and the other fingers are spread around the thoracic cage and angled toward the body's side to create a consistent, compressive force across the thoracic cage. The subject is then asked to breathe in deeply and breathe out. While breathing out, rhythmic oscillatory compression in the posterior and caudal direction is applied to the chest wall. By the end of the expiratory phase, the compressive force is maintained, and the subject is asked to take another deep breath. In this way, the subject encountered some resistance equivalent to the chest-wall movement during inspiration. The maneuver is repeated for five respiratory cycles, after that the therapist slowly reduces the compressive force and withdraws his hands.
  Arms: Thoracic lymphatic pump technique
Other: Exercises (stretching and strenghtening ) — stretching exercises include: Hamstring stretching exercises
  Lower back stretching exercises :
  strenghtening exercises include:
  Abdominal curl up exercises :
  Supine bridging exercises. Trunk extension exercises

SUMMARY:
The purpose of the study is to compare between the combined effect of thoracic lymphatic pump technique with exercises and exercises alone on pain intensity using Visual Analogue Scale (VAS), lumbar spine mobility using Modified-Modified Schober test (MMST) and functional disability level using Oswestary Disability Index (ODI) on patients with CMLBP.

DETAILED DESCRIPTION:
Study design: This study will be randomizaed controlled trail.1. Participants:forty-two patients with chronic mechanical low back pain. age:20-45. Th sample size population: was calculated using the G*power program 3.1.9 (G power program version 3.1, Heinrich-Heine-University, Düsseldorf, Germany) for one tailed test. Sample size calculation based on F tests (ANOVA: Special effects and interactions), Type I error (a) = 0.05, power (1-ß error probability) = 0.80, Pillai V = 0.3300000 and effect size f (V) = 0.8 with 2 independent groups comparison for 3 major variable outcomes. The appropriate minimum sample size for this study was 42 patients (21 patients in each group). Procedure:First, the purpose of the study will be explained to the patients and the procedures are fully explained. Then, patients will be asked to participate in the study. If they accepted, an informed consent form will be signed and randomly assigned in one of two groups (by closed envelope method). All subjects will be evaluated for their pain intensity,lumbar spine mobility and functional disability level. All patients will be tested before and after the treatment program (12 treatment sessions, 3 sessions per week for 4 weeks). Each patient will receive exercises (stretching and strengthening exercises) for the control group (A), the stretching exercises include (Hamstring stretching- Lower back stretching) and the strengthening exercises- include (Abdominal curl up- Supine bridging-Trunk extension). For the experimental group (B), they will receive exercises (stretching and strengthening exercises) then the thoracic lymphatic pump technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients (both genders) with a chief complain of Chronic mechanical low back pain without leg pain (Al Sulaimy et al., 2018).
* Age of the patient 20- 45 years old (Al Sulaimy et al., 2018).
* Pain more than three months

Exclusion Criteria:

* Patient with Spondylolysis (Steele et al., 2016).
* Patient with tumor, infection (Ulger et al., 2017).
* Patient with cauda equina syndrome who need urgent surgery (Ulger et al., 2017).
* Patients with previous lumber surgery (Amundsen et al., 2018).
* Patient with Deep venous thrombosis (DVT) (Alves et al., 2020).
* Patient with Congestive heart failure (Alves et al., 2020).
* Patient with Renal failure (Forner-Cordero et al., 2021).
* Patient with uncontrolled hypertension (Forner-Cordero et al., 2021).

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  Arabic version of the Visual analogue scale (VAS) will be used, the subject will mark on a 0-10 graphic rating scale in which the (0) value indicating no pain, and (10) indicating the most severe pain experienced. Then a ruler will be used to measure the distance from zero, the recorded number will be rounded to the closest value

SECONDARY OUTCOMES:
Functional disability level | 4 weeks
  Functional disability level will be assessed by Oswestary disability index (ODI) which is a clinical assessment tool that provides an estimate of disability expressed as a percentage score. It consists of ten sections that assess pain, personal care, lifting, walking, sitting, standing, sleeping, sexual life, social life and travelling. It consists of ten multiple choice questions for back pain; patient selects one sentence out of six of the best describes her/his pain. High scores indicate great pain (Nishant et al., 2014). Arabic version of the questionnaire will be used and the questions are going to be explained to the subjects. For illiterate subjects, the therapist will read and explain the questions for them

OTHER OUTCOMES:
Lumbar spine mobility | 4 weeks
  Modified-Modified Schober test (MMST) which is a valid and reliable tool, is used to assess lumbar spine mobility through flexion, extension movements

CONTACTS AND LOCATIONS:
Locations (1):
- Basma Hesham, Giza, Egypt